CLINICAL TRIAL: NCT03061357
Title: Incorporating Wearable Technology Into Physical Activity Instructional Program: A Cluster Randomized Trial in University Settings
Brief Title: Physical Activity Intervention Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Youngdeok Kim, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 505314
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Physical Activity
Keywords: activity tracker; behavior change
MeSH Terms: conditions — Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Participant
Masking Description: All participants in both intervention and control arms were not disclosed to the specific purpose of the study in order to prevent the subject-expectancy effects on study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity tracker group (Experimental): Participants in intervention arm were provided with a small and lightweight activity tracker, Misfit Flash (Misfit Wearables Co., Burlingame, CA), that can be worn with a clasp or watch band. A handout detailing the step-by-step instructions for utilizing the activity tracker with Misfit App on their smartphone was provided. There was no intervention component mandated in the curriculum of intervention PAIP courses; rather, participants were continuously encouraged by the instructors to track their activity levels and use all the features in Misfit App on a daily basis as they learned health benefits of PA and as to how to develop individualized, life-long PA plan during the course of semester.
  Interventions: Behavioral: Activity tracker
- Control group (No Intervention): Participants in control arm did not receive any additional instructions other than the scheduled class activities based on the standardized core-curriculum of PAIP

INTERVENTIONS:
Behavioral: Activity tracker — Misfit Flash (Misfit Wearables Co., Burlingame, CA) activity tracker
  Arms: Activity tracker group

SUMMARY:
This project was to examine the effects of incorporating modern wearable technology into the credit-based Physical Activity Instructional Program for promoting habitual levels of physical activity among college students.

DETAILED DESCRIPTION:
This project was a cluster randomized trial examining the effects of utilizing a wearable activity tracker in a credit-based Physical Activity Instructional Program on promoting habitual levels of physical activity (PA) in college students.

The project was conducted in a large public university located in the mid-south region of the US. The university offers more than one hundred 1-credit hour PAIPs per academic semester. Considering the pilot nature of the study, the target PAIPs was limited to those meeting the following inclusion criteria: 1) PAIP with a size of 30 students that generally show an approximately equal gender distribution; and 2) PAIP that delivers the principles and practice of individually tailored habitual activity plans. The investigators randomly selected 14 eligible PAIPs and assigned them into intervention (k=7) and control (k=7) groups. The outcome measures of interests were the changes in objectively and subjectively measured physical activity over an academic semester.

ELIGIBILITY:
Inclusion Criteria:

* healthy college students who were enrolled in 1-credit physical activity instruction programs.

Exclusion Criteria:

* did not wish to participate;
* have currently used their own wearable activity tracker;
* indicated any major physical, psychiatric, or cardiovascular-related problems diagnosed by a physician.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in objectively measured physical activity to 15 weeks | baseline and 15 weeks
  Physical activity was objectively measured using an ActiGraph Actitrainer (ActiGraph LLC, Pensacola, FL, USA) accelerometer.

SECONDARY OUTCOMES:
Change from baseline in subjectively measured physical activity | baseline and 15 weeks
  Physical activity was subjectively measured using International Physical Activity Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Youngdeok Kim, PhD, Principal Investigator — Texas Tech University

IPD SHARING:
Plan to Share IPD: No